CLINICAL TRIAL: NCT04703582
Title: Relationship Between Morbimortality and Basal Activated Clotting Time (ACT) in Patients Undergoing Vascular Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TCA-2020-92
Record Dates: First submitted 2021-01-04; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Artery Disease, Peripheral; Aortic Diseases; Carotid Artery Diseases; Other Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Aortic Diseases; Carotid Artery Diseases; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Activated clotting time — Relationship between elongated baseline activated clotting time and comorbidity

SUMMARY:
Check whether patients with higher comorbidity and risk of complication, estimated using the V (p) -POSSUM score, ACS NSQIP and the ASA classification, present higher baseline activated clotting time values.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing vascular surgery requiring intraoperative heparinization

Exclusion Criteria:

* Pregnant women
* SARS-CoV-2 PCR positive (performed 24-72h prior to surgery)
* Severe plaquetopenia <50,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing vascular surgery consecutively in the first semester of 2021, for a period of one month, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change on baseline Activated Clotting Time with comorbidities | 1 day - surgery day
  Activted Clotting Time will be measured with Haemocron Machine just before surgery. Comorbidities will be measured with V(p)Possum, AC NSQUIP and ASA scales.